CLINICAL TRIAL: NCT01188304
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Effect of 150 µg Aleglitazar Once Daily in Healthy Subjects Treated With 325 mg Aspirin Once Daily on Renal Function, Renin-angiotensin System and Platelet Aggregation
Brief Title: A Study of Aleglitazar in Combination With Aspirin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP25329
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aleglitazar; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: aleglitazar; Drug: aspirin
- 2 (Placebo Comparator)
  Interventions: Drug: aspirin; Drug: placebo

INTERVENTIONS:
Drug: aleglitazar — repeated daily doses
  Arms: 1
Drug: aspirin — repeated daily doses
Drug: placebo — repeated daily doses
  Arms: 2

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group study will investigate the safety and tolerability, and the effect of aleglitazar in combination with aspirin on renal function, renin-angiotensin system and platelet aggregation in healthy volunteers. Volunteers will be randomized to receive daily doses of aleglitazar or placebo in combination with aspirin. The anticipated time on study drug is 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, aged 40 to 65 years inclusive
* Body Mass Index (BMI) between 18 and 35 kg/m2 inclusive
* Females of child-bearing potential must be willing to use two acceptable methods of contraception during the study and at least 3 months before start of the study
* Non-smoker or currently smoking less than 5 cigarettes (or equivalent amount of other tobacco products) per day and is willing and able to stop smoking during the period in study center
* Volunteer drinks no more than 3 cups of coffee, tea or soft drinks per day and is willing and able to stop drinking coffee, tea and soft drinks during the period in study center

Exclusion Criteria:

* Any clinically relevant abnormal laboratory test results at screening
* Volunteer has taken any prescribed, herbal or over-the-counter medication within 2 weeks prior to first dosing
* A history of any clinical significant gastro-intestinal, cardiovascular, musculoskeletal, endocrine, hematological, psychiatric, renal, hepatic, bronchopulmonary or neurological conditions or lipid disorders
* A positive test for human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B or hepatitis C
* History of intolerance to non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin, history of gastric or duodenal ulceration, personal or family history of abnormal clotting or bleeding

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of aleglitazar in combination with aspirin on measured glomerular filtration rate | 13 weeks

SECONDARY OUTCOMES:
To investigate the effect of aleglitazar in combination with aspirin on renal plasma flow, filtration fraction and estimated glomerular filtration rate | 13 weeks
To investigate the effect of aleglitazar in combination with aspirin on renin-angiotensin system and on anti-diuretic hormone | 13 weeks
To investigate the effect of aspirin in combination with aleglitazar on platelet function and serum thromboxane B2 | 13 weeks
To investigate the pharmacokinetics of aleglitazar when co-administered with aspirin | 13 weeks
To investigate safety and tolerability of aleglitazar | 13 weeks
To investigate the effect of aleglitazar in combination with aspirin on electrolytes and osmolality clearances | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- San Antonio, Texas, United States